CLINICAL TRIAL: NCT00070421
Title: @neWorld: A Virtual Community For Kids With Cancer
Brief Title: Study of @neWorld: A Virtual Community for Children With Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Leap of Faith Technologies (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Other Study IDs: LFT-NEWORLD; CDR0000334398 (Registry Identifier: PDQ (Physician Data Query)); WCCC-2000-194
Record Dates: First submitted 2003-10-03; First posted 2003-10-07 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2004-12

CONDITIONS: Leukemia; Lymphoma; Psychosocial Effects of Cancer and Its Treatment; Unspecified Childhood Solid Tumor, Protocol Specific
Keywords: psychosocial effects of cancer and its treatment; unspecified childhood solid tumor, protocol specific; childhood acute lymphoblastic leukemia in remission; childhood acute myeloid leukemia in remission; recurrent childhood acute lymphoblastic leukemia; recurrent childhood acute myeloid leukemia; recurrent childhood large cell lymphoma; recurrent childhood lymphoblastic lymphoma; recurrent childhood small noncleaved cell lymphoma; stage I childhood Hodgkin lymphoma; stage I childhood large cell lymphoma; stage I childhood lymphoblastic lymphoma; stage I childhood small noncleaved cell lymphoma; stage II childhood Hodgkin lymphoma; stage II childhood large cell lymphoma; stage II childhood lymphoblastic lymphoma; stage II childhood small noncleaved cell lymphoma; stage III childhood Hodgkin lymphoma; stage III childhood large cell lymphoma; stage III childhood lymphoblastic lymphoma; stage III childhood small noncleaved cell lymphoma; stage IV childhood Hodgkin lymphoma; stage IV childhood large cell lymphoma; stage IV childhood lymphoblastic lymphoma; stage IV childhood small noncleaved cell lymphoma; recurrent/refractory childhood Hodgkin lymphoma
MeSH Terms: conditions — Leukemia; Lymphoma; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Dendritic Cell Sarcoma, Interdigitating; Burkitt Lymphoma; Recurrence | interventions — Psychiatric Rehabilitation

INTERVENTIONS:
Procedure: complementary or alternative medicine procedure
Procedure: management of therapy complications
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Using an Internet Web site that enables children with cancer to interact online with classmates, participate in classroom activities, get easy-to-read medical information, and chat with family members, medical staff, and other children with cancer may help children cope with isolation, fear, and decreased self-esteem.

PURPOSE: This phase I/II trial is studying the effectiveness of an Internet Web site in providing social support and education to children who are undergoing treatment for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Develop an Internet-based application that allows pediatric patients with cancer to enter a virtual community with the following capabilities:

  * Interact with classmates and participate in classroom activities via e-mail, chat groups, online field trips, art studio, music room, and game room
  * Identify and interact with a community of peers with similar medical conditions
  * Access a dictionary to get medical information in understandable terms
  * Interact with the medical community online
  * Interact with family members online
* Determine the acceptability of this program among groups of these patients and their classmates, teachers, family members, and healthcare providers using focus groups.
* Determine the effect of this program on self-esteem, coping behaviors, perceived social support, cancer-relevant medical knowledge, and feelings of control over health destiny in these patients.
* Determine the effect of this program on the performance of these patients in school.
* Determine the effect of this program in alleviating psychological distress in these patients.

OUTLINE: This is a multicenter study.

* Phase I: Students, family members, teachers, and health providers participate in focus groups to provide system design and implementation input and to assess overall acceptability of a prototype Internet-based application for pediatric cancer patients.
* Phase II: Patients are assigned to 1 of 2 groups, based on participating center.

  * Group 1: Patients have access to and utilize the Internet-based application @neWorld.
  * Group 2: Patients do not have access to or utilize @neWorld. In both groups, patients complete questionnaires measuring psychological distress, quality of life, self-esteem, coping behaviors, perceived academic and social competence, perceived social support, cancer-relevant medical knowledge, feelings of control over health destiny, utilization of psychological services, and performance in school at baseline and 3 and 6 months.

PROJECTED ACCRUAL: A total of 94 patients (44 for group 1 and 50 for group 2) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of cancer
* Currently receiving treatment for cancer

PATIENT CHARACTERISTICS:

Age

* 10 to 15

Performance status

* Active

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Able to read and speak English

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Dates: Start 2003-04; Study Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barbara Rapchak, Study Chair — Leap of Faith Technologies
Locations (1):
- Leap of Faith Technologies, Incorporated, Crystal Lake, Illinois, United States